CLINICAL TRIAL: NCT00200018
Title: ASSIST: Appetite Suppression Induced by Stimulation Trial
Brief Title: Study of Weight Loss Using Gastric Stimulation in Obese Patients With Type 2 Diabetes
Acronym: ASSIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Kristin Schwartz, Medtronic Neuromodulation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1163-85585
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: Severe to Morbid Obesity and Type 2 Diabetes
Keywords: Obesity; Morbid obesity; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Obesity, Morbid; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Enterra Therapy System (H9900014)

SUMMARY:
The purpose of this study is to test the effect of an implanted device that stimulates the stomach on weight loss in patients suffering from obesity and type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes with HbA1c of 7.5 - 11%
* Willing to make behavior and lifestyle modifications
* No previous bariatric surgery (gastric bypass, gastric banding)
* Meet additional study criteria

Exclusion Criteria:

* History of substance abuse or chemical dependency with in the last 3 years
* Prior GI surgery for morbid obesity or any gastric surgery for conditions other than obesity or diabetes
* Severe congestive heart failure
* Any underlying illness other than diabetes or obesity that affects gastrointestinal motility
* Currently taking medications for weight loss

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2005-06; Primary Completion 2007-02 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Mean excess weight loss and percent excess weight loss | 12 months

SECONDARY OUTCOMES:
Diabetes status and use of diabetes medication | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: ASSIST Team, Study Chair — Medtronic
Locations (2):
- United States (2):
  - La Jolla, California
  - Eagan, Minnesota